CLINICAL TRIAL: NCT05833438
Title: A Single-arm, Pilot Study of Venetoclax in Combination with 5 Days Azacitidine in Treatment-naïve Subjects with Acute Myelogenous Leukemia Who Are ≥18 Years of Age and Not Eligible for Standard Induction Therapy (VENAZA-5S PILOT TRIAL)
Brief Title: Venetoclax in Combination with 5 Days Azacitidine in Untreated AML Patients, Not Eligible for Standard Induction Therapy
Acronym: VENAZA-5S
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: AbbVie (Industry); University Hospital Leipzig, Hematology Diagnostics Laboratory (Unknown); University of Leipzig, Clinical Trial Centre (ZKS) (Unknown)
Responsible Party: Principal Investigator, Klaus Metzeler, Prof. Dr. med. Klaus Metzeler, University of Leipzig
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VENAZA-5S; 2022-501537-23-00 (Other: EU CT Number (EMA,CTIS ))
Record Dates: First submitted 2023-03-04; First posted 2023-04-27 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Venclyxto; Venetoclax; Azacitidine; Hematologic Diseases; Acute Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VEN+AZA-5 (Experimental): Azacitidine (AZA) 75 mg/m2, d1-5 of each 28 day cycle (SC) in combination with Venetoclax (VEN): 400 mg daily (orally)
  Interventions: Drug: VEN+AZA-5

INTERVENTIONS:
Drug: VEN+AZA-5 — Up to 6 cycles: Azacitidine (AZA) 75 mg/m2, d1-5 of each 28 day cycle (SC) in combination with Venetoclax (VEN): 400 mg daily (orally)

SUMMARY:
Acute myeloid leukemia (AML): continuous oral Venetoclax (VEN) and 7 days of s.c. Azacitidine (AZA) per 28-day cycle = standard of care for intensive induction therapy ineligible AML patients in Germany

The VENAZA-5S pilot trial: AZA administration reduced to 5 days within each cycle to improve tolerability and treatment adherence due to less neutropenic infections, less treatment interruptions and less hospitalizations.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a uniformly fatal disease if untreated. The combination of continuous oral Venetoclax (VEN) and 7 days of s.c. Azacitidine (AZA) per 28-day cycle has recently emerged as the new standard of care for AML patient who are ineligible for intensive induction therapy, and has been widely adopted in Germany.

The VENAZA-5S pilot trial aims to reduce the reported hematological toxicity profile of this currently approved combination, while preserving efficacy, by modifying AZA administration to 5 days within each cycle. The hypothesis is that this modification will not interfere with the response rates achieved by the combination, but will rather improve tolerability and treatment adherence due to less neutropenic infections, less treatment interruptions and hospitalizations, and thus result in better quality of life and favorable long-term outcomes in elderly or comorbid AML patients. This single-arm pilot study is intended to generate first data on the efficacy and toxicity of 5 days AZA + VEN, which will be compared to a historical control cohort treated with the current standard of 7 days AZA + VEN.

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed diagnosis of AML by World Health Organization (WHO) criteria 2016
* Ineligible for treatment with a standard cytarabine and anthracycline induction regimen due to age or comorbidities
* Age ≥ 18 years
* Life expectancy of at least 12 weeks

Key Exclusion Criteria:

* Prior treatment for AML or myelodysplastic syndrome (MDS) with one of the following:

  * Hypomethylating agent (HMA)
  * Chemotherapeutic agent
  * Chimeric Antigen Receptor (CAR)-T cell therapy
  * Experimental therapies
  * Note: Prior use of hydroxyurea is allowed
* History of myeloproliferative neoplasm (MPN)
* Diagnosis of acute promyelocytic leukemia (APL)
* Presence of favorable-risk karyotype abnormalities: t(15;17), t(8;21), inv(16) or t(16;16)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the response rate defined as the rate of CR/CRi after up to 6 cycles of therapy (best response). | best response after up to 6 cycles (each cycle is 28 days)
  Bone marrow assessments will be performed at least at screening, at the end of cycle 1, after cycle 4 and after cycle 6 resp. end of treatment (EOT). Criteria for disease status / response assessment follow the ELN-2022 recommendations .

SECONDARY OUTCOMES:
Rate of CR or CRi by the Initiation of Cycle 2 | At the end of Cycle 1 (each cycle is 28 days)
  Rate of CR or CRi by the Initiation of Cycle 2. Criteria for disease status / response assessment follow the European LeukemiaNet (ELN) - 2022 recommendations.
Rate of CR with partial hematologic recovery (CRh) after up to 6 cycles of therapy | after up to 6 cycles (each cycle is 28 days)
  Rate of CR with partial hematologic recovery (CRh) after up to 6 cycles of therapy. Criteria for disease status / response assessment follow the ELN-2022 recommendations.
Time from initiation of treatment (C1D1) until achievement of CR or CRi | from start of treatment (C1D1) until up to 6 cycles (each cycle is 28 days)
  Time from initiation of treatment (C1D1) until achievement of CR or CRi. Criteria for disease status / response assessment follow the ELN-2022 recommendations.
Objective response rate | at EOT, after up to 6 cycles therapy (each cycle is 28 days)
  Objective response rate (CR, CRh, CRi, MLFS). Criteria for disease status / response assessment follow the ELN-2022 recommendations.
Event free survival (EFS) | From start of treatment to the date of relapse from CR or CRi, treatment failure (i.e., no CR or CRi after up to 6 cycles (each cycle is 28 days) of therapy or disease progression requiring treatment discontinuation), or death from any cause.
  Event free survival (EFS), defined as the number of days from start of treatment to the date of relapse from CR or CRi, treatment failure (i.e., no CR or CRi after 6 cycles (each cycle is 28 days) of therapy or disease progression requiring treatment discontinuation), or death from any cause.
Overall survival (OS) | From start of treatment to date of death from any cause. OS will be assessed until 3 months after end of treatment of the last patient on study.
  Overall survival (OS), defined as the number of days from start of treatment to death from any cause.
  After EOT, patients will be further followed up for survival until the end of the trial is reached (= last patient out, i.e. when the last surviving patient has reached the 3-month follow-up visit after EOT). Therefore, the duration of follow-up can differ between patients but is at least 3 months after EOT.
Descriptive assessment of measurable residual disease (MRD) levels on study treatment, determined by quantitative PCR or targeted next-generation sequencing | From Screening until EOT (after up to 6 cycles (each cycle is 28 days))
  Determined by quantitative PCR or targeted next-generation sequencing. Molecular profiling and MRD assessment of all patients will be carried out centrally (Hämatologisches Diagnostiklabor, Universitätsklinikum Leipzig), at least at screening, at the end of cycle 1, after cycle 4 and after cycle 6 resp. end of treatment (EOT).
Time to treatment discontinuation | From start of treatment to day of treatment discontinuation (within up to 6 cycles (each cycle is 28 days))
  Time to treatment discontinuation, defined as the number of days from start of treatment to premature stop of treatment. The stop date is the date the first cycle that was not given should have started as scheduled. This endpoint will be analyzed with death and progression or relapse as competing risk.
Rate of patients with at least one treatment interruption | From start of treatment until EOT (after up to 6 cycles (each cycle is 28 days))
  Rate of patients with at least one treatment interruption, i.e. a delay of the next cycle, and duration of treatment interruptions.
Delay of subsequent cycles, dose reductions or shortening/interruption of study drug administration | From start of treatment until EOT (after up to 6 cycles (each cycle is 28 days))
  Delay of subsequent cycles, dose reductions or shortening/interruption of study drug administration
Duration of patient hospitalization | From start of treatment until EOT (after up to 6 cycles (each cycle is 28 days))
  Duration of patient hospitalization, defined as days in hospital from start of treatment until EOT.
Quality of life (QoL) | From Screening until EOT (after up to 6 cycles (each cycle is 28 days))
  The established cancer-specific Core Quality of Life questionnaire QLQ-C30 from the EORTC (European Organisation for Research) will be used for QoL measurement, at screening and at the beginning of each cycle and at EOT.

OTHER OUTCOMES:
Incidence of Adverse Events [Safety and Tolerability] | From start of treatment until 35±7 days after EOT
  Descriptive analysis of adverse events for all patients having received at least one dose of investigational medicinal product (IMP). Adverse events will be documented from day 1 of the first treatment cycle until 35±7 days after EOT.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Metzeler, Prof. Dr., Principal Investigator — Universitätsklinikum Leipzig, Klinik und Poliklinik für Hämatologie, Zelltherapie und Hämostaseologie
Locations (10):
- Germany (10):
  - Helios Klinikum Berlin-Buch Klinik für Hämatologie und Stammzelltransplantation, Berlin
  - Klinikum Chemnitz gGmbH Klinik für lnnere Medizin Ill, Chemnitz
  - Carl-Thiem-Klinikum Cottbus gGmbH, Cottbus
  - Universitatsklinikum Carl Gustav Carus Dresden an der TU Dresden Medizinische Klinik und Poliklinik 1 Bereich Hamatologie, Dresden
  - Universitätsklinikum Heidelberg, Innere Medizin V; Klinik für Hämatologie, Onkologie und Rheumatologie, Heidelberg
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Hämatologie, Zelltherapie und Hämostaseologie, Leipzig
  - Kliniken Maria Hilf GmbH, Klinik für Hämatologie, Onkologie und Gastroenterologie, Mönchengladbach
  - Rotkreuzklinikum München, III. Medizinische Abteilung, München
  - Klinikum rechts der lsar der TU München, Klinik und Poliklinik für lnnere Medizin Ill, München
  - Kliniken Sindelfingen,Medizinische Klinik I, Sindelfingen

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of this study, after deidentification
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 3 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal for individual participant data meta-analysis.